CLINICAL TRIAL: NCT04356378
Title: Long Term Physical Functional Performance in Daily Living in SARS-CoV2 Infected Patients Hospitalized in the Acute Phase Then Requiring Rehabilitation: a Multicentric Observational Study
Brief Title: Long Term Physical Functional Limitations in Daily Living in SARS-CoV2 Infected Patients Hospitalized in the Acute Phase Then Requiring Rehabilitation
Acronym: CAPACoV19
Status: Completed | Type: Observational
Sponsor: CHU de Reims (Other)
Responsible Party: Sponsor
Other Study IDs: PO20055
Record Dates: First submitted 2020-04-17; First posted 2020-04-22 (Actual); Last update posted 2024-06-04 (Actual); Status verified 2024-06

CONDITIONS: Infection With Coronavirus SARS-CoV2
Keywords: observational study; cohort study; coronavirus infections; respiratory distress syndrome; adult; rehabilitation; physical functional performance; long term care; exercise tolerance; clinical study
MeSH Terms: conditions — Coronavirus Infections; Respiratory Distress Syndrome | interventions — Electronic Health Records

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- "infection with coronavirus SARS-CoV2" group: "SARS-CoV2 infected patients" group: in-patient in the acute phase then requiring rehabilitation.
  Interventions: Other: Data record

INTERVENTIONS:
Other: Data record — Data record

SUMMARY:
Infection with coronavirus SARS-CoV2 (COVID-19 disease) is unique with its speed of propagation, structural medical reorganizations and length of stay in intensive care needed, diversity of the affected population (in particular between young persons or fragile subjects), and impact on physical and mental health generated by confinement of populations.

Fatigue is a major component of COVID-19. Global muscular weakness is related to immobility, inflammation, corticosteroids treatment, hypoxemia due to pulmonary and/or cardiac infectious attacks and undernutrition suggests major physical functional repercussions. Thus, patients affected by COVID-19 with acute hospital management require sometimes complex rehabilitation management.

Retrospective studies on physical functional capacities in patients infected with SARS CoV1 showed long term physical activity limitations.

DETAILED DESCRIPTION:
The aim of this study is to study factors associated with physical functional limitations in daily living in patients SARS-CoV2 infected and hospitalized in the acute phase then requiring rehabilitation.

ELIGIBILITY:
Inclusion criteria :

* patient infected with SARS-CoV2
* in-patient hospitalization in the acute phase because SARS-CoV2 infection
* patient requiring rehabilitation after SARS-CoV2 infection acute phase
* patient adult, aged more than 18 years old
* patient accepting to participate in the study

Exclusion criteria :

* patient with cognitive disorder (Folstein Mini-Mental State Examination less than 22 on 30 points)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: SARS-CoV2 infected patients, hospitalized in the acute phase then requiring rehabilitation follow-up.
Sampling Method: Non-Probability Sample
Enrollment: 149 (Actual)
Dates: Start 2020-06-02 (Actual); Primary Completion 2021-08-20 (Actual); Study Completion 2022-01-20 (Actual)

PRIMARY OUTCOMES:
Physical functional limitations | 12 months
  Physical functional limitations evaluated using 'sit to stand' test. The patient, seated in a chair without armrest, his arms crossed over his shoulders, should get up and sit down without help of the upper limbs as many times as possible in one minute.

CONTACTS AND LOCATIONS:
Locations (1):
- Damien JOLLY, Reims, France